CLINICAL TRIAL: NCT04022213
Title: Phase II Combination of 131I-Omburtamab Radioimmunotherapy and External Beam Radiotherapy for Desmoplastic Small Round Cell Tumor
Brief Title: A Study of the Drug I131-Omburtamab in People With Desmoplastic Small Round Cell Tumors and Other Solid Tumors in the Peritoneum
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-182
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Desmoplastic Small Round Cell Tumor; Peritoneal Cancer; Peritoneal Carcinoma
Keywords: Solid Tumor; Peritoneal Solid Tumor; DSRC; I131-Omburtamab; Memorial Sloan Kettering Cancer Center; 19-182
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Participants with DSRCT who have undergone GTR of their abdominopelvic disease and who have no definitive radiological evidence of disease in liver or outside the abd/pelvis. Patients if deemed of likely benefit to the patient after completing IP RIT plus WAP-IMRT, or will be mandated if ANC is persistently <500/ul despite use of G-CSF for >1 week, or if patients experience life threatening febrile neutropenia.
  Interventions: Drug: 131 I-omburtamab; Radiation: WAP-IMRT
- Group B (Experimental): DSRCT patients who have macroscopic residual disease OR who have previously experienced progression of disease while on treatment but have subsequently had a GTR
  Interventions: Drug: 131 I-omburtamab
- Group C (Experimental): Participants with tumors other than DSRCT and will be enrolled onto an assessment arm to determine eligibility. Immunohistochemistry to assess B7H3 expression will be performed on frozen or paraffin embedded tissue using omburtamab (frozen tissue) or a commercially available anti-B7H3 antibody (if paraffin embedded).
  Interventions: Drug: 131 I-omburtamab

INTERVENTIONS:
Drug: 131 I-omburtamab — Single dose of IP RIT administered through an IP catheter with 131 I-omburtamab at 80mCi/m2
Radiation: WAP-IMRT — Group A participants will receive WAP-IMRT approximately 2-4 weeks after completing IP RIT. A dose of 30 Gy will be delivered in 20 fractions of 1.5 Gy given once daily, 5 days per week over the course of approximately 4 weeks
  Other Names: Intensity Modulated Radiation Therapy
  Arms: Group A

SUMMARY:
The purpose of this study is to test any good and bad effects of the study drug 131I-omburtamab. 131I-omburtamab could prevent the cancer from returning, or delay the cancer from getting worse, but it could also cause side effects. Researchers hope to learn more about how 131I-omburtamab works in the body, and how effective it is in treating cancer. 131I-Omburtamab is not approved by the FDA to treat DSRCT or other cancers of the peritoneum.

ELIGIBILITY:
Inclusion Criteria:

* Have the diagnosis of DSRCT confirmed at MSKCC
* Age >1 year and able to cooperate with radiation safety restrictions during therapy period.
* Prior to intraperitoneal catheter placement

  * At least 1 weeks must have elapsed since prior chemotherapy
  * At least 2 weeks must have elapsed since biologic therapy
  * Toxicities of prior therapy must have resolved to grade 1 or less or to the patient's baseline

At the completion of surgery, patients must fulfill all of the additional following criteria:

* Have no definitive radiological evidence of disease active in liver or outside the abdomen/pelvic OR have had GTR of this disease at the time of catheter placement

Exclusion Criteria:

* Prior progression of disease
* Prior hypothermic intraperitoneal chemotherapy (HIPEC)
* Cardiac, pulmonary, and neurologic toxicities are greater grade 1 per NCI CTCAE version 5
* Renal, gastrointestinal, and hepatic, toxicities are greater than grade 2 (per NCI CTCAE version 5)
* History of allergy to mouse proteins
* Patients with grade 4 hypersensitivity reaction to radiolabeled iodine

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival/PFS | Up to 2 years after treatment is discontinued
  Progression free survival after RIT + WA-IMRT.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Slotkin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org